CLINICAL TRIAL: NCT06725537
Title: Comprehensive Demographics and Clinical Profile of NSCLC Patients: Analyzing Treatment Patterns With PD-L1 Stratification
Brief Title: Comprehensive Demographics and Clinical Profile of NSCLC Patients
Acronym: CA209-1529
Status: Not yet recruiting | Type: Observational
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1529
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer Non Small Cell
Keywords: neoplasia; lung; metastasis; first line treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Advances in the treatment of non-small cell lung cancer in the last decade have been significant. Currently, there are several first-line therapeutic options. The molecular biology of the disease, biomarkers and the patient's clinical characteristics can assist in decision making. The study in question aims to retrospectively evaluate the patterns of choice in the first line treatment of metastatic non-small cell lung cancer without driver mutations, from 2019 to 2022 in 7 centers in Brazil.

DETAILED DESCRIPTION:
Lung cancer is the most incident neoplasm in the world (considering both sexes), with 2.4 million (12.4%) new cases per year, based on estimates from the Global Cancer Observatory (Globocan) in 2022 (1). Non-small cell histology (NSCLC) is the most common and represents around 76% of lung cancer cases (2). Despite improvements in its prevention and diagnosis, a large proportion of patients are diagnosed in the advanced stage of the disease (57%) (3) and some of those diagnosed with localized disease will experience recurrence of the neoplasm. In this sense, choosing the most appropriate first-line treatment is necessary.

The last decade has been marked by advances in the treatment of lung cancer. Regarding metastatic non-small cell lung cancer without target mutation, the inclusion of immunotherapy in the therapeutic arsenal has led to a significant increase in survival rates (2). Currently, with the exception of a few patients given specific contraindications, an immunological check point inhibitor (ICI) will be present in the first-line treatment of this group (4). The current challenge is choosing the best treatment approach for each patient.

The use of ICI in the first line can be used as monotherapy or combination therapy. In 2016, the KEYNOTE-024 study was published in NEJM, a pioneer in this scenario, which evaluated the use of Pembrolizumab monotherapy in patients with a TPS score ≥50% (5). It was a positive study for its primary outcome of progression-free survival (PFS), with a median PFS of 10.3 months for the group that received Immunotherapy versus 6.7 months for the group that received chemotherapy (CT) (HR 0.5; 0.37 - 0.68 ). It also demonstrated a significant gain in overall survival (OS), with 5-year follow-up reaffirmation - median OS 26.3 months for Pembrolizumab versus 13.4 months for CT (HR 0.62; 0.48 - 0.81) (6). Five years after first publication of KN-024, the EMPOWER Lung-01 study was published in the Lancet (7). He evaluated the use of Cemiplimab in the same population and also obtained positive results in relation to OS (26.1 months ICI arm versus 13.3 months in the CT arm - HR 0.57; 0.46 - 0.71) (8) and PFS.

In relation to patients with low expression (1-49%) or without PD-L1 expression (negative), the combination of immunotherapy and chemotherapy appears to be a good treatment strategy. The KEYNOTE-189 study, published in NEJM in 2018, evaluated the use of Pembrolizumab associated with doublet chemotherapy (Carboplatin or Cisplatin + Pemetrexed) in patients with lung adenocarcinoma without target alteration (EGFR or ALK) regardless of PD-L1 expression (9). Their results show a survival benefit with the use of the combination with ICI and updated data on 5-year OS maintain this gain (19.4% versus 11.3%) (10). In the same year, the KEYNOTE-407 study evaluated the use of Pembrolizumab in combination with CT in patients with squamous histology. Similarly, it demonstrated a survival benefit (11). In its most recent update, the 5-year OS data maintains benefit for the ICI combination arm, with a 29% reduction in the risk of death (12).

In this same subgroup, other medications were evaluated. The IMPOWER-150 study evaluated the use of Atezolizumab in combination with CT, with and without the VEFG inhibitor (Bevacizumab) (13). It included patients with metastatic lung adenocarcinoma and included patients with EGFR and ALK mutations, but only in a small proportion. The study met its coprimary endpoints of PFS and OS, with a median OS of 19.0 months for the ICI+CT+Bevacizumab combination versus 14.7 months for the CT+Bevacizumab arm (14).

Finally, the ICI combination was also evaluated. Three studies are worth highlighting. The first of them, CheckMate-227, evaluated the use of Ipilimumab and Nivolumab, without the addition of CT (15). There was an OS benefit from the combination, regardless of PD-L1 expression, with 6-year OS of 22% in the PD-L1 positive population and 16% in the negative one (16). The second, CheckMate-9LA evaluated the use of Ipilimumab and Nivolumab, associated with two CT cycles. The scheme led to a benefit in OS, with a reduction in the risk of death by 27% in five-year data update (17). Similarly, the POSEIDON study evaluated the use of Durvalumab and Tremelimumab associated with CT, leading to a benefit in OS from the combination (18).

When confronted with numerous options, oncologists seek unique characteristics and biomarkers to inform their decisions. They consider patient factors such as age, comorbidities, and performance status. Regarding tumor patterns, details like histology, the location of metastatic disease (CNS vs. non-CNS), and PD-L1 expression are also crucial in guiding their choices.

In relation to patients with actionable target mutations, standard first-line management may differ from that previously explored. Therefore, it is extremely important to investigate molecular biology, especially in non-squamous histology and in non-smoking patients. The evaluation of the EGFR and ALK genes is essential, as well as the BRAF, RAS, RET, MET, NTRK, HER2 and ROS1 genes.

In the current scenario, there are several treatment options targeting specific actionable mutations approved in Brazil. Testing for these key mutations is widely available, and assessing the quality, reliability, and turnaround time of the test, as well as the molecular alterations considered by the physician when choosing the first line and sequencing the treatment, is important.

In summary first-line treatment of NSCLC has peculiarities and molecular evaluation is mandatory. Several treatment regimens have demonstrated benefit in OS, but they have not been directly compared (15). Given the options presented, the current challenge is choosing the best treatment approach for each patient (16). The search for biomarkers that predict response, which help in decision making, is tireless. Currently, this definition is made by specialist oncologists, who use the data presented so far to make the choice. Subgroup assessments in each study, the toxicity profile and dosage are points taken into consideration. Thus, the identification of data that assists doctors in this decision-making becomes attractive.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Histological diagnosis of advanced non-small cell cancer;
* Clinical and demographic data available in medical records;

Exclusion Criteria:

* Patients with localized disease that can be treated locally;
* Non-epithelial histology;
* small cell carcinoma
* neuroendocrine tumor

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a histological diagnosis of advanced non-small cell lung cancer, over 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
treatment regimen decision option one | In 30 days
  immunotherapy versus chemotherapy, this outcome will be evaluated based on data from medical records and available laboratory results
treatment regimen decision option two | In 30 days
  dual immunotherapy, this outcome will be evaluated based on data from medical records and available laboratory results

SECONDARY OUTCOMES:
Survival analysis | In 24 months
  Survival will be analyzed secondarily, using the variable time to death

CONTACTS AND LOCATIONS:
Overall Officials: Sofia V Mendes, MD, Principal Investigator — Instituto D'Or de Pesquisa e Ensino

IPD SHARING:
Plan to Share IPD: No